CLINICAL TRIAL: NCT06772506
Title: Clinical and Patient-centered Outcomes After Minimally Invasive Non-surgical Therapy for the Treatment of Splinted Stage IV Periodontitis - Randomized Controlled Clinical Trial
Brief Title: Minimally Invasive Non-surgical Therapy for the Treatment of Splinted Stage IV Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, shaimaa hamdy, lecturer in department of periodontology, Nahda University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MINST in Periodontitis; 2019-002239-27 (EudraCT Number)
Record Dates: First submitted 2025-01-03; First posted 2025-01-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Periodontitis; Stage IV Periodontitis; Minimally Invasive Treatment; Splints
Keywords: periodontitis; stage IV; MINST; splint
MeSH Terms: conditions — Periodontitis | interventions — Listerine; Ethanol; methyl salicylate; Menthol; Thymol; Splints

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- conventional periodontal treatment with ultrasonic device and manual instruments (Experimental): conventional non-surgical techniques with ultrasonic and manual scaler instruments
  Interventions: Procedure: Non Surgical Periodontal Treatment includes post operative mouth wash with Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%)
- Placebo minimally invasive non surgical technique with mini five and after five instruments (Placebo Comparator): and minimally invasive non-surgical technique using mini five and after five instruments+ ultrasonic device for supragingival instrumentation
  Interventions: Procedure: Minimally invasive non-surgical technique with mini five and after five minimally invasive instrument plus splint

INTERVENTIONS:
Procedure: Non Surgical Periodontal Treatment includes post operative mouth wash with Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%) — non-surgical technique plus splint and ultrasonic device with 200 mg Tetracycline
  Arms: conventional periodontal treatment with ultrasonic device and manual instruments
Procedure: Minimally invasive non-surgical technique with mini five and after five minimally invasive instrument plus splint — minimally invasive instruments, with mini five and after five minimally invasive instrument ultrasonic scaler device, conventional radiographic device and periodontal instruments with post-operative 1 gram penicillin for 3 days regulatory Statement: This study does not include an FDA-regulated device intervention, as the tools utilized are not the subject of investigation but are instead employed as part of routine clinical
  Other Names: with ultrasonic device; mini five and after five instruments
  Arms: Placebo minimally invasive non surgical technique with mini five and after five instruments

SUMMARY:
Conventional periodontal treatment typically involves a combination of non-surgical and surgical approaches, such as scaling and root planing, followed by flap surgery and guided tissue regeneration. While these methods have demonstrated some success in managing periodontal disease, the low success rate in complex cases has prompted the exploration of alternative treatment modalities. One such approach is minimally invasive, non-surgical monotherapy, which aims to address the etiological source of the inflammation without the need for invasive surgical intervention.

Guided tissue regeneration, a well-established technique in periodontal treatment, employs physical barrier membranes to exclude the proliferation of unwanted gingival fibroblasts and allow the regeneration of tooth-supporting structures such as the alveolar bone, periodontal ligament, and cementum.

Recent advancements in dental therapies have led to the exploration of minimally invasive non-surgical approaches that aim to achieve comparable outcomes with reduced morbidity. This protocol outlines a randomized clinical trial to evaluate the efficacy and safety of a minimally invasive non-surgical monotherapy in treating patients with stage 4 periodontitis.

Is minimally invasive non-surgical technique more effective in reducing tooth mobility and improving clinical parameters than conventional non-surgical technique?

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease that affects the supporting structures of the teeth, including the gingiva, periodontal ligament, cementum, and alveolar bone. The advanced stages of periodontitis, such as stage 4, are characterized by severe tissue destruction, deepened pocket depths, and alveolar bone loss, which can ultimately lead to tooth mobility, drifting, and loss. Effective therapeutic interventions are necessary to halt the progression of the disease and potentially regenerate the lost periodontal tissues.

Conventional periodontal treatment typically involves a combination of non-surgical and surgical approaches, such as scaling and root planing, followed by flap surgery and guided tissue regeneration. While these methods have demonstrated some success in managing periodontal disease, the low success rate in complex cases has prompted the exploration of alternative treatment modalities. One such approach is minimally invasive, non-surgical monotherapy, which aims to address the etiological source of the inflammation without the need for invasive surgical intervention.

Guided tissue regeneration, a well-established technique in periodontal treatment, employs physical barrier membranes to exclude the proliferation of unwanted gingival fibroblasts and allow the regeneration of tooth-supporting structures such as the alveolar bone, periodontal ligament, and cementum.

Recent advancements in dental therapies have led to the exploration of minimally invasive non-surgical approaches that aim to achieve comparable outcomes with reduced morbidity. This protocol outlines a randomized clinical trial to evaluate the efficacy and safety of a minimally invasive non-surgical monotherapy in treating patients with stage 4 periodontitis.

Is minimally invasive non-surgical technique more effective in reducing tooth mobility and improving clinical parameters than conventional non-surgical technique?

ELIGIBILITY:
Inclusion Criteria:

* periodontitis stage III and IV
* Mobility grade 2
* age from 18-55 years
* medically free
* nonsmoker
* Single-rooted teeth

Exclusion Criteria:

* Medically compromised patient
* smokers
* Bad oral hygiene
* Non-surgical or surgical periodontal treatment in the past 12months.
* Prolonged treatment with antibiotics or anti-inflammatory agents within 6months before periodontal therapy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 18-55 year old
Enrollment: 40 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
CAL by millimeters | baseline, 3months and 6 months
  Clinical attachment loss

CONTACTS AND LOCATIONS:
Locations (1):
- Egypt, Cairo, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
after publishing, i will share it